CLINICAL TRIAL: NCT06029855
Title: Effects Of Kabat Rehabilitation Versus Mime Therapy On Facial Disability And Synkinesis In Patients Of Bell's Palsy
Brief Title: Kabat Rehabilitation Versus Mime Therapy on Facial Disability and Synkinesis in Patients of Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-406-05-2023
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-01

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; Kabat Rehabilitation; Mime Therapy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kabat Therapy (Active Comparator): Kabat exercises primarily assist functional response in defective muscles through the general structure of muscles experiencing resistance. After 6th week, resting and voluntary symmetries were recorded.
  Interventions: Other: Kabat Therapy
- Mime Therapy (Experimental): Mime therapy utilizes emotional input to access better movement patterns. It is beneficial as it improves circulation and maintains muscle properties.
  Interventions: Other: Mime Therapy

INTERVENTIONS:
Other: Kabat Therapy — The participants of group A will receive Kabat Rehabilitation with routine physical therapy. The protocol will be given to the participants for three sessions/week for six weeks. Each session will be of 30 minutes.
  Arms: Kabat Therapy
Other: Mime Therapy — The participants of group B will receive Mime Therapy in addition to routine physical therapy. The protocol will be given to the participants once a week for six weeks, while physical therapy will be given on alternate days. Each session will be of 30 minutes.
  Arms: Mime Therapy

SUMMARY:
Bell's palsy, also called idiopathic facial paralysis, is a common cause of unilateral facial paralysis. It is one of the most common neurological disorders of the cranial nerves.

DETAILED DESCRIPTION:
Bell's palsy is an alarming condition of rapid onset, which paralyzes half of the facial muscles. Kabat rehabilitation is a manual resistance technique that promotes a basic pattern of movement through facilitation, inhibition, and resistance of a group of muscles. It increases the functioning and power of facial muscles while Mime therapy results in immediate improvement of function and integrity of facial muscles. It also mitigates synkinesis in Bell's palsy. Both techniques are easy to apply. They are clinically important techniques that are easily understood by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 25-50 years.
2. Both male and female.
3. Unilateral bell's paralysis.
4. Not congenital in origin.
5. Sub-acute and chronic cases.

Exclusion Criteria:

1. Other neurological deficits include epilepsy and Alzheimer's disease.
2. Traumatic onset.
3. Surgical reconstruction (nerve or muscle reconstruction).
4. Mental and psychological disorders i.e., schizophrenia, bipolar disorders.
5. Skin diseases (eczema, urticarial) as electrical stimulation may affect the results.
6. Any contraindications for massage like sunburn, bruising, or cuts.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Synkinesis | It will be assessed at baseline, at the third week and at six week.
  Synkinesis will be accessed through the "House-Brackmann Scale". It is classified as a universal scale. This scale analyses the symmetry, synkinesis, stiffness, and global mobility of the face. It is divided into six categories (normal, mild dysfunction, moderate dysfunction, moderately severe dysfunction, severe dysfunction, and total paralysis) and is a 0-6-point scale with 6 representing total paralysis.
Level of Facial Disability | Change in functional status will be measured at the baseline, at 3rd week and at 6th week.
  The level of Facial disability will be measured through the "Facial Disability Index Scale". This scale has ten items that evaluate the patient's physical and social aspects (mastication, deglutition, communication, labial mobility, emotional alterations, and social integration). It uses a hundred-point scale with a higher score indicating less impairment. 24 Minimum score for physical functioning: 0, Maximum score for physical functioning: 25, Minimum score for social and well-being: 5, Maximum score for social and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Dr Ahmed, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Immediately after publication

REFERENCES:
- [Derived] Amjad A, Jamil A, Fatima N, Javaid HB, Zahid H. Effects of Kabat rehabilitation versus mime therapy on facial disability and synkinesis in patients of Bell's palsy. J Pak Med Assoc. 2024 Nov;74(11):1927-1931. doi: 10.47391/JPMA.11247. PMID 39548608